CLINICAL TRIAL: NCT00560950
Title: A Multicenter, Open-Label Study of the Safety, Tolerability, and Immunogenicity of Revaccination With PNEUMOVAX(TM) 23 Vaccine (Pneumococcal Vaccine Polyvalent, Merck & Co., Inc.) in Older Adults
Brief Title: Revaccination With PNEUMOVAX(TM) 23 in Older Adults (V110-007)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V110-007; 2007_540
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Results first posted 2009-05-25 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-03

CONDITIONS: Pneumococcal Infection
MeSH Terms: conditions — Pneumococcal Infections | interventions — 2,4,5,4'-tetrachlorodiphenylsulfoxide; Pneumococcal Vaccines

ARMS (2):
- 1st Revaccination Group (Experimental)
  Interventions: Biological: pneumococcal 23v polysaccharide vaccine
- 2nd Revaccination Group (Experimental)
  Interventions: Biological: pneumococcal 23v polysaccharide vaccine

INTERVENTIONS:
Biological: pneumococcal 23v polysaccharide vaccine — Duration of Treatment: Single vaccination on Day 1
  Other Names: V110; PNEUMOVAX

SUMMARY:
The purpose of this study is to determine that revaccination of Pneumococcal Vaccine is well tolerated and produces an immune response in older adults.

DETAILED DESCRIPTION:
This study is an extension study (V110-007-10) which met requirements for posting on clinicaltrials.gov. The original study (V110-007-00) was completed in 2004 and did not meet the criteria for registration.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal or negative urine pregnancy test if female
* No fever on the day of vaccination

Exclusion Criteria:

* History of allergy to vaccine components
* History of pneumococcal disease
* Received any live virus vaccination within 4 weeks prior to study start
* Received any inactivated vaccination within 7 days prior to study start
* Received any blood products within 5 months prior to study start
* Participated in an investigational drug or vaccine study in the past 30 days
* Received immunosuppressive therapy
* Patient has an immune deficiency

Min Age: 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2007-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Musher DM, Manoff SB, McFetridge RD, Liss CL, Marchese RD, Raab J, Rueda AM, Walker ML, Hoover PA. Antibody persistence ten years after first and second doses of 23-valent pneumococcal polysaccharide vaccine, and immunogenicity and safety of second and third doses in older adults. Hum Vaccin. 2011 Sep;7(9):919-28. doi: 10.4161/hv.7.9.15996. Epub 2011 Sep 1. PMID 21860256
- [Result] Manoff SB, Liss C, Caulfield MJ, Marchese RD, Silber J, Boslego J, Romero-Steiner S, Rajam G, Glass NE, Whitney CG, Carlone GM. Revaccination with a 23-valent pneumococcal polysaccharide vaccine induces elevated and persistent functional antibody responses in adults aged 65 > or = years. J Infect Dis. 2010 Feb 15;201(4):525-33. doi: 10.1086/651131. PMID 20088694

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase III study. The first patient was enrolled (FPE) on 13-Jul-2007. The last patient last visit (LPLV) was on 30-May-2008. A total of 5 US study centers were involved in the recruitment.
Pre-assignment Details: Base trial 4/97-4/98 Prior to results posted Initial: subjects received 1st or 2nd dose of PN23 Persistence: followed immune response 5 yrs; ended 4/03 Extension 7/07-4/08: enrolled 9-10 yrs after base. 1dose of PN23 Blood drawn Days 1&30, immune response to 8 serotypes measured 143 of 400 enrolled: difficulty enrolling eligible/interested subjects
Groups:
- 1st Revaccination Group: Received primary vaccination with Pneumovax 23 during the initial phase and 1st revaccination in the extension phase
- 2nd Revaccination Group: Received 1st revaccination with Pneumovax 23 during the initial phase and 2nd revaccination in the extension phase
Period: Overall Study
Arm/Group | 1st Revaccination Group | 2nd Revaccination Group
Started | 72 | 71
Completed | 71 | 71
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1st Revaccination Group | 2nd Revaccination Group | Total
Number analyzed (Participants) | 72 | 71 | 143
Age, Continuous [Mean (Full Range); unit: years] | 74.6 [60 to 93] | 77.1 [60 to 88] | 75.8 [60 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 45 | 90
  Male | 27 | 26 | 53

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Concentration for Prevaccination (Day 1) to Postvaccination (Day 30) During the Extension Phase Subjects Completing the Extension for Serotype 3
Description: Blood drawn at Day 1 and Day 30 of the extension study were used to measure IgG antibody levels to 8 pneumococcal polysaccharide serotypes (3, 4, 6B,8, 9V, 12F, 14, 23F) by ELISA.
Time Frame: Day 1 & Day 30
Population: All eligible participants
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units/mL
Arm/Group | 1st Revaccination Group Day 1 | 1st Revaccination Group Day 30 | 2nd Revaccination Group Day 1 | 2nd Revaccination Group Day 30
Number analyzed (Participants) | 68 | 67 | 67 | 67
gpELISA units/mL | 0.6 [0.5 to 0.8] | 1.4 [1.1 to 1.8] | 0.7 [0.5 to 0.8] | 1.2 [0.9 to 1.6]

2. Primary Outcome: Geometric Mean Concentration for Prevaccination (Day 1) to Postvaccination (Day 30) During the Extension Phase Subjects Completing the Extension for Serotype 4
Description: Blood drawn at Day 1 and Day 30 of the extension study were used to measure IgG antibody levels to 8 pneumococcal polysaccharide serotypes (3, 4, 6B, 8, 9V, 12F, 14, 23F) by ELISA.
Time Frame: Day 1 & Day 30
Population: All eligible participants
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units/mL
Arm/Group | 1st Revaccination Group Day 1 | 1st Revaccination Group Day 30 | 2nd Revaccination Group Day 1 | 2nd Revaccination Group Day 30
Number analyzed (Participants) | 68 | 67 | 67 | 67
gpELISA units/mL | 1.1 [0.8 to 1.5] | 3.0 [2.2 to 3.9] | 1.7 [1.4 to 2.2] | 3.0 [2.2 to 4.0]

3. Primary Outcome: Geometric Mean Concentration for Prevaccination (Day 1) to Postvaccination (Day 30) During the Extension Phase Subjects Completing the Extension for Serotype 6B
Description: as for outcome 2
Time Frame: Day 1 & Day 30
Population: All eligible participants
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units/mL
Arm/Group | 1st Revaccination Group Day 1 | 1st Revaccination Group Day 30 | 2nd Revaccination Group Day 1 | 2nd Revaccination Group Day 30
Number analyzed (Participants) | 68 | 67 | 67 | 67
gpELISA units/mL | 2.0 [1.5 to 2.7] | 4.6 [3.3 to 6.4] | 3.0 [2.2 to 4.2] | 5.2 [3.6 to 7.5]

4. Primary Outcome: Geometric Mean Concentration for Prevaccination (Day 1) to Postvaccination (Day 30) During the Extension Phase Subjects Completing the Extension for Serotype 8
Description: as for outcome 2
Time Frame: Day 1 & Day 30
Population: All eligible participants
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units/mL
Arm/Group | 1st Revaccination Group Day 1 | 1st Revaccination Group Day 30 | 2nd Revaccination Group Day 1 | 2nd Revaccination Group Day 30
Number analyzed (Participants) | 68 | 67 | 67 | 67
gpELISA units/mL | 3.0 [2.4 to 3.7] | 9.3 [7.4 to 11.8] | 3.4 [2.7 to 4.4] | 7.4 [5.8 to 9.3]

5. Primary Outcome: Geometric Mean Concentration for Prevaccination (Day 1) to Postvaccination (Day 30) During the Extension Phase Subjects Completing the Extension for Serotype 9V
Description: as for outcome 2
Time Frame: Day 1 & Day 30
Population: All eligible participants
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units/mL
Arm/Group | 1st Revaccination Group Day 1 | 1st Revaccination Group Day 30 | 2nd Revaccination Group Day 1 | 2nd Revaccination Group Day 30
Number analyzed (Participants) | 68 | 67 | 67 | 67
gpELISA units/mL | 2.7 [2.0 to 3.6] | 7.2 [5.7 to 9.1] | 4.1 [3.2 to 5.4] | 8.0 [6.0 to 10.7]

6. Primary Outcome: Geometric Mean Concentration for Prevaccination (Day 1) to Postvaccination (Day 30) During the Extension Phase Subjects Completing the Extension for Serotype 12F
Description: as for outcome 2
Time Frame: Day 1 & Day 30
Population: All eligible participants
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units/mL
Arm/Group | 1st Revaccination Group Day 1 | 1st Revaccination Group Day 30 | 2nd Revaccination Group Day 1 | 2nd Revaccination Group Day 30
Number analyzed (Participants) | 68 | 67 | 67 | 67
gpELISA units/mL | 0.4 [0.3 to 0.6] | 1.5 [1.0 to 2.1] | 0.8 [0.6 to 1.2] | 1.5 [1.0 to 2.2]

7. Primary Outcome: Geometric Mean Concentration for Prevaccination (Day 1) to Postvaccination (Day 30) During the Extension Phase Subjects Completing the Extension for Serotype 14
Description: as for outcome 2
Time Frame: Day 1 & Day 30
Population: All eligible participants
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units/mL
Arm/Group | 1st Revaccination Group Day 1 | 1st Revaccination Group Day 30 | 2nd Revaccination Group Day 1 | 2nd Revaccination Group Day 30
Number analyzed (Participants) | 68 | 67 | 67 | 67
gpELISA units/mL | 9.2 [6.9 to 12.2] | 18.0 [13.4 to 24.0] | 10.3 [8.2 to 13.0] | 17.2 [13.3 to 22.2]

8. Primary Outcome: Geometric Mean Concentration for Prevaccination (Day 1) to Postvaccination (Day 30) During the Extension Phase Subjects Completing the Extension for Serotype 23F
Description: as for outcome 2
Time Frame: Day 1 & Day 30
Population: All eligible participants
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units/mL
Arm/Group | 1st Revaccination Group Day 1 | 1st Revaccination Group Day 30 | 2nd Revaccination Group Day 1 | 2nd Revaccination Group Day 30
Number analyzed (Participants) | 68 | 67 | 67 | 67
gpELISA units/mL | 1.8 [1.2 to 2.6] | 4.7 [3.1 to 7.1] | 2.8 [2.0 to 3.8] | 5.6 [3.8 to 8.2]

ADVERSE EVENTS:
Arm/Group | 1st Revaccination Group | 2nd Revaccination Group
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/71
Other Adverse Events (participants affected / at risk) | 48 | 60
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | 1st Revaccination Group | 2nd Revaccination Group
Lymphadenopathy (Blood and lymphatic system disorders) | 0/71 | 1/71
Dry Eye (Eye disorders) | 0/71 | 1/71
Lacrimation Increased (Eye disorders) | 1/71 | 0/71
Macular Degeneration (Eye disorders) | 0/71 | 1/71
Abdominal Pain Upper (Gastrointestinal disorders) | 0/71 | 1/71
Aphthous (Gastrointestinal disorders) | 1/71 | 0/71
Diarrhoea (Gastrointestinal disorders) | 0/71 | 1/71
Nausea (Gastrointestinal disorders) | 0/71 | 3/71
Oral Disorder (Gastrointestinal disorders) | 1/71 | 0/71
Anaesthesia (General disorders) | 0/71 | 1/71
Chills (General disorders) | 1/71 | 7/71
Coldness (General disorders) | 0/71 | 1/71
Erythema (General disorders) | 14/71 | 21/71
Fatigue (General disorders) | 18/71 | 27/71
Induration (General disorders) | 0/71 | 1/71
Oedema Peripheral (General disorders) | 2/71 | 0/71
Pain (General disorders) | 18/71 | 24/71
Pain (Injection site) (General disorders) | 44/71 | 53/71
Paraesthesia (General disorders) | 0/71 | 1/71
Peripheral Coldness (General disorders) | 0/71 | 1/71
Pruritus (General disorders) | 2/71 | 4/71
Pyrexia (General disorders) | 1/71 | 4/71
Swelling (General disorders) | 14/71 | 28/71
Warmth (General disorders) | 2/71 | 1/71
Cystitis (Infections and infestations) | 1/71 | 0/71
Nasopharyngitis (Infections and infestations) | 0/71 | 1/71
Procedural Pain (Injury, poisoning and procedural complications) | 0/71 | 1/71
Blood Pressure Increased (Investigations) | 0/71 | 1/71
Hyperglycaemia (Metabolism and nutrition disorders) | 0/71 | 1/71
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0/71 | 1/71
Back Pain (Musculoskeletal and connective tissue disorders) | 2/71 | 1/71
Joint Range of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1/71 | 0/71
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0/71 | 2/71
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 2/71 | 1/71
Neck Pain (Musculoskeletal and connective tissue disorders) | 0/71 | 1/71
Headache (Nervous system disorders) | 13/71 | 18/71
Hypoaesthesia (Nervous system disorders) | 1/71 | 0/71
Migrane (Nervous system disorders) | 0/71 | 1/71
Disorientation (Psychiatric disorders) | 0/71 | 1/71
Insomnia (Psychiatric disorders) | 1/71 | 0/71
Restlessness (Psychiatric disorders) | 1/71 | 0/71
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1/71 | 0/71
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 0/71 | 1/71

LIMITATIONS AND CAVEATS:
Open-label non-randomized group of subjects enrolled in this extension. Subjects recruited from original study which completed five years previously.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.